CLINICAL TRIAL: NCT07144631
Title: PENS-P: Peroneal Electrical Nerve Stimulation in Pregnancy for Restless Legs Syndrome (RLS)
Brief Title: Peroneal Electrical Nerve Stimulation in Pregnancy for Restless Legs Syndrome
Acronym: PENS-P
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: American College of Chest Physicians (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2313348
Record Dates: First submitted 2025-08-11; First posted 2025-08-27 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Restless Leg Disorder; Restless Leg Syndrome (RLS); Pregnancy; Sleep Disorder (Disorder)
Keywords: Restless Legs Syndrome; Pregnancy; Sleep Disorders in Pregnancy; Maternal Sleep Health; Peroneal Nerve Stimulation; Neuromodulation
MeSH Terms: conditions — Restless Legs Syndrome; Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: All enrolled participants will receive the same intervention (TOMAC™ peroneal nerve stimulation).
  There is no randomization to different arms or a control/placebo group in this pilot study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- TOMAC™ Peroneal Nerve Stimulation (Experimental): Participants will receive TOMAC™ peroneal nerve stimulation (PNS) therapy for Restless Legs Syndrome (RLS) during pregnancy. Following a supervised in-clinic titration session with uterine contraction and fetal monitoring at ≥28 weeks' gestation, participants will use the device at home for 8 weeks. Each therapy session lasts 30 minutes and can be performed as many times as needed daily, prioritizing periods of high symptom burden or before bedtime. Outcomes include feasibility, acceptability, adherence and maternal-fetal safety.
  Interventions: Device: Peroneal Nerve Stimulation (PNS) Device

INTERVENTIONS:
Device: Peroneal Nerve Stimulation (PNS) Device — The TOMAC™ system is a non-invasive, wearable peroneal nerve stimulator that delivers high-frequency electrical stimulation to the common peroneal nerves at the fibular head. It is FDA-cleared for the treatment of moderate-to-severe Restless Legs Syndrome (RLS) in adults but has not been studied in pregnancy. In this trial, pregnant participants will undergo an in-clinic titration session with uterine contraction and fetal monitoring at ≥28 weeks' gestation to determine comfortable therapeutic intensity. They will then use the device at home for 8 weeks, up to four 30-minute sessions daily, prioritizing periods of high symptom burden or before bedtime. Outcomes will assess feasibility, acceptability, adherence, symptom improvement, sleep quality, and maternal-fetal safety.

SUMMARY:
The goal of this study is to evaluate whether peroneal electrical nerve stimulation (PNS) using the TOMAC™ device is a feasible, acceptable, and safe non-pharmacologic intervention for managing Restless Legs Syndrome (RLS) during pregnancy. This pilot study will also collect preliminary information on symptom relief, sleep quality, and maternal-fetal safety associated with device use.

The main questions the study aims to answer are:

Is TOMAC™ PNS a feasible and acceptable intervention for RLS in pregnant individuals? Are there any maternal, fetal, or neonatal safety concerns with PNS use during pregnancy? What are the patterns of adherence, tolerance, and usability of the TOMAC™ device in this population?

Participants will:

Use a non-invasive TOMAC™ peroneal nerve stimulator during 30-minute sessions as needed, for 8 weeks.

Complete questionnaires assessing feasibility, acceptability, symptom severity, and sleep quality (including AIM, IAM, FIM, IRLS, PGI-I, PSQI, ESS, FOSQ, and MOS-II).

Wear an actigraphy monitor to collect objective sleep data at baseline and at 4 weeks.

Attend scheduled follow-up visits and phone check-ins for maternal vital signs, uterine contraction and fetal monitoring, and neonatal outcome assessment.

This is a prospective, open-label, single-arm pilot study enrolling 15 pregnant participants between 21 and 26 weeks' gestation. Findings will provide the first dataset on the feasibility, acceptability, and safety of TOMAC™ PNS in pregnancy and inform the design of a future randomized controlled trial.

DETAILED DESCRIPTION:
This is a prospective, open-label, single-arm pilot study designed to assess the feasibility, acceptability, and preliminary safety of TOMAC™ peroneal electrical nerve stimulation (PNS) for the treatment of Restless Legs Syndrome (RLS) during pregnancy.

RLS affects approximately 20-30% of pregnant individuals, with symptoms often worsening during the second and third trimesters. It is associated with disrupted sleep, decreased quality of life, and adverse pregnancy outcomes such as gestational hypertension, preeclampsia, prolonged labor, and increased cesarean delivery rates. Pharmacologic therapies for RLS are generally avoided during pregnancy because of limited data on fetal safety, highlighting the need for effective, non-pharmacologic alternatives.

The TOMAC™ system is a non-invasive, wearable, high-frequency peroneal nerve stimulator that delivers bilateral stimulation to the common peroneal nerves. It is FDA De Novo granted for use in adults with moderate to severe RLS but has not been evaluated in pregnant populations. Safety rationale for this study is informed by evidence from other neuromodulation therapies, such as sacral nerve stimulation, which have been used safely during pregnancy without observed maternal or fetal harm.

Primary objectives are to evaluate the feasibility and acceptability of TOMAC™ PNS using validated implementation measures, including the Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), and Feasibility of Intervention Measure (FIM).

Secondary objectives include assessment of adherence, dose tolerance, usability, maternal and fetal safety, and exploratory evaluation of symptom improvement and sleep quality through the International Restless Legs Syndrome Rating Scale (IRLS), Patient Global Impression of Improvement (PGI-I), Pittsburgh Sleep Quality Index (PSQI), Epworth Sleepiness Scale (ESS), Functional Outcomes of Sleep Questionnaire (FOSQ), and Medical Outcomes Study Sleep Problem Index II (MOS-II).

Fifteen pregnant individuals between 21 and 26 weeks of gestation with a confirmed diagnosis of RLS will be enrolled. Following baseline assessments, participants will undergo an in-person titration session under clinical supervision, which includes uterine contraction and fetal monitoring performed at ≥28 weeks' gestation to ensure maternal and fetal safety.

Participants will then use the TOMAC™ device at home for an 8-week intervention, performing self-administered 30-minute sessions as needed, preferably during periods of symptom distress or prior to sleep.

Data will be collected from patient-reported outcomes, actigraphy sleep recordings, device usage logs, and maternal-fetal safety monitoring. Follow-up includes biweekly phone check-ins, an in-person mid-study visit at week 4, a final in-person visit at week 8, and a three-month postpartum safety follow-up.

This pilot study will generate the first prospective data on the feasibility, acceptability, and safety of peroneal nerve stimulation in pregnancy, providing foundational evidence for future randomized controlled trials evaluating TOMAC™ PNS as a pregnancy-safe, non-pharmacologic treatment for RLS and its potential to improve maternal sleep and pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Pregnant individuals between 21 and 26 weeks' gestation at enrollment
* Singleton pregnancy without known fetal anomalies
* Confirmed clinical diagnosis of Restless Legs Syndrome (RLS) according to International Restless Legs Syndrome Study Group (IRLSSG) criteria, confirmed by a sleep medicine specialist to exclude RLS mimics
* Able and willing to provide informed consent
* Able and willing to comply with study procedures, including device usage, questionnaires, adherence diaries, and follow-up assessments up to 3 months postpartum

Exclusion Criteria:

Pregnancy-related:

* History of preterm labor
* Known fetal anomalies identified prior to enrollment

Neurological and neuromuscular disorders:

* Pre-existing neuromuscular disorders affecting balance or gait
* Severe peripheral neuropathy involving the lower legs
* Epilepsy or history of seizures

Cardiovascular and circulatory conditions:

* History of deep vein thrombosis (DVT)
* Circulatory conditions contraindicating peroneal nerve stimulation (PNS) device use

Dermatological conditions:

* Skin conditions at device application sites
* Known allergy to device materials

Other sleep disorders:

• Inadequately treated severe primary sleep disorders other than RLS (e.g., untreated severe sleep apnea, severe insomnia unrelated to RLS)

Device and treatment experience exclusions (based on RESTFUL trial criteria):

* Prior use of the study device or any neurostimulation device for RLS treatment
* Presence of active medical implants (e.g., pacemakers, spinal cord stimulators)

Other medical conditions:

* Participants undergoing dialysis treatment
* Severe psychiatric conditions (e.g., bipolar disorder, psychosis, severe anxiety or depression) that may interfere with adherence or accurate symptom reporting
* Any condition deemed by investigators to pose safety risks or impede participation

Other exclusions:

* Unable or unwilling to operate the device safely and independently
* Unable to participate reliably in follow-up assessments or complete self-reported diaries

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Intervention Measure (AIM) Score | Baseline to 8 weeks of intervention
  The Acceptability of Intervention Measure (AIM) is a validated 4-item questionnaire assessing participants' perceptions of how acceptable the intervention is. Scores range from 1 to 5. Higher scores indicate greater acceptability.
Intervention Appropriateness Measure (IAM) Score | Baseline and Week 8 of intervention
  The Intervention Appropriateness Measure (IAM) is a validated 4-item questionnaire assessing participants' perceptions of how appropriate the intervention is for their condition. Scores range from 1 to 5. Higher scores indicate greater appropriateness.
Feasibility of Intervention Measure (FIM) Score | Baseline and Week 8 of intervention
  The Feasibility of Intervention Measure (FIM) is a validated 4-item questionnaire assessing participants' perceptions of how feasible it is to use the intervention. Scores range from 1 to 5. Higher scores indicate greater feasibility.

SECONDARY OUTCOMES:
Adherence to Maximum Allowed Device Sessions | Throughout 8 weeks of intervention
  Adherence will be measured as the proportion of actual device sessions used compared to the maximum allowed use (as many as needed 30-minute sessions for 8 weeks). Data will be collected from device logs and participant diaries. Results will be reported as the percentage of completed sessions relative to the maximum allowable sessions.
Mean Session Duration | Continuous during 8-week intervention
  Average duration of each stimulation session, recorded by device logs. Results will be reported in minutes per session.
Mean Stimulation Voltage Used During Device Sessions | Continuous during 8-week intervention
  Average stimulation voltage delivered by the peroneal nerve stimulation (PNS) device during participant sessions, recorded from device logs. Results will be reported as mean voltage across all sessions.
Number of Participants With Treatment-Related Adverse Events (AEs) | Throughout 8-week intervention
  Number of participants experiencing treatment-emergent adverse events related to device use, as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Results will be reported as total number of participants.
Number of Participants With Serious Adverse Events (SAEs) | Throughout 8-week intervention
  Number of participants experiencing serious adverse events related to device use, as assessed by CTCAE v4.0. Results will be reported as total number of participants.
Change in Maternal Systolic Blood Pressure | Baseline, Week 4, Week 8
  Maternal systolic blood pressure measured at in-clinic visits using automated sphygmomanometer. Results will be reported as mean change in millimeters of mercury (mmHg).
Change in Maternal Diastolic Blood Pressure | Baseline, Week 4, Week 8
  Maternal diastolic blood pressure measured at in-clinic visits using automated sphygmomanometer. Results will be reported as mean change in millimeters of mercury (mmHg).
Change in Maternal Heart Rate | Baseline, Week 4, Week 8
  Maternal heart rate measured at in-clinic visits using automated sphygmomanometer. Results will be reported as mean change in beats per minute (bpm).
Incidence of Uterine Irritability During Titration | At ≥28 weeks of pregnancy during titration session
  Proportion of participants who experience uterine irritability during the in-clinic titration session (≥28 weeks gestation). Uterine irritability is defined per protocol as ≥10 contractions within a 20-minute period, measured using external tocodynamometry. Results will be reported as percentage of participants.
Incidence of Fetal Distress During Titration | At ≥28 weeks of pregnancy during titration session
  Proportion of participants who experience fetal distress during the in-clinic titration session (≥28 weeks gestation). Fetal distress is defined as one or more of the following:
  * FHR bradycardia <110 bpm for ≥10 minutes
  * FHR tachycardia >160 bpm for ≥10 minutes
  * Minimal/absent variability (<5 bpm amplitude for ≥20 minutes)
  * Recurrent decelerations (≥3 late or variable decelerations in 20 minutes)
  Results will be reported as percentage of participants.
Incidence of Uterine Irritability Associated With Fetal Distress | At ≥28 weeks of pregnancy during titration session
  Proportion of participants who experience both uterine irritability (≥10 contractions in 20 minutes) and concurrent fetal distress during the same titration session, as defined above. Results will be reported as percentage of participants.
Infant Birth Weight | At delivery
  Infant birth weight measured at delivery. Results will be reported in grams.
Neonatal Apgar Score at 1 Minute | At delivery (1 minute)
  Neonatal Apgar score assessed at 1 minute after delivery. Scores range from 0 to 10, with higher scores indicating better neonatal condition. Results will be reported as mean score.
Neonatal Apgar Score at 5 Minutes | At delivery (5 minutes)
  Neonatal Apgar score assessed at 5 minute after delivery. Scores range from 0 to 10, with higher scores indicating better neonatal condition. Results will be reported as mean score.
Neonatal Health Outcomes at 3 Months Postpartum | 3 months postpartum
  Proportion of infants with adverse health outcomes, including but not limited to growth restriction, feeding difficulties, recurrent hospitalizations, or clinician-diagnosed developmental concerns. Outcomes will be reported as percentage of infants, based on maternal report confirmed by pediatric/OB medical records.

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study is a small pilot with a limited sample size and data will only be used for the purposes outlined in the approved protocol. The IRB-approved consent form does not include provisions for external data sharing.

REFERENCES:
- [Background] Yoshimura C, Arima H, Amagase H, Takewaka M, Nakashima K, Imaoka C, Miyanaga N, Obama H, Fujita M, Ando SI. Idiopathic and secondary restless legs syndrome during pregnancy in Japan: Prevalence, clinical features and delivery-related outcomes. PLoS One. 2021 May 11;16(5):e0251298. doi: 10.1371/journal.pone.0251298. eCollection 2021. PMID 33974646
- [Background] Yaiesh SM, Al-Terki AE, Al-Shaiji TF. Safety of Sacral Nerve Stimulation in Pregnancy: A Literature Review. Neuromodulation. 2016 Oct;19(7):770-779. doi: 10.1111/ner.12450. Epub 2016 Jun 10. PMID 27286484
- [Background] Winkelman JW, Berkowski JA, DelRosso LM, Koo BB, Scharf MT, Sharon D, Zak RS, Kazmi U, Falck-Ytter Y, Shelgikar AV, Trotti LM, Walters AS. Treatment of restless legs syndrome and periodic limb movement disorder: an American Academy of Sleep Medicine clinical practice guideline. J Clin Sleep Med. 2025 Jan 1;21(1):137-152. doi: 10.5664/jcsm.11390. PMID 39324694
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Walters AS, LeBrocq C, Dhar A, Hening W, Rosen R, Allen RP, Trenkwalder C; International Restless Legs Syndrome Study Group. Validation of the International Restless Legs Syndrome Study Group rating scale for restless legs syndrome. Sleep Med. 2003 Mar;4(2):121-32. doi: 10.1016/s1389-9457(02)00258-7. PMID 14592342
- [Background] Vahdat M, Sariri E, Miri S, Rohani M, Kashanian M, Sabet A, Zamani B. Prevalence and associated features of restless legs syndrome in a population of Iranian women during pregnancy. Int J Gynaecol Obstet. 2013 Oct;123(1):46-9. doi: 10.1016/j.ijgo.2013.04.023. Epub 2013 Jul 22. PMID 23886452
- [Background] Teresi JA, Yu X, Stewart AL, Hays RD. Guidelines for Designing and Evaluating Feasibility Pilot Studies. Med Care. 2022 Jan 1;60(1):95-103. doi: 10.1097/MLR.0000000000001664. PMID 34812790
- [Background] Szymanski JK, Slabuszewska-Jozwiak A, Jakiel G. Sacral Neuromodulation in Pregnant Women-A Case Report and Literature Review. Int J Environ Res Public Health. 2022 Jul 8;19(14):8340. doi: 10.3390/ijerph19148340. PMID 35886191
- [Background] Steinweg K, Nippita T, Cistulli PA, Bin YS. Maternal and neonatal outcomes associated with restless legs syndrome in pregnancy: A systematic review. Sleep Med Rev. 2020 Dec;54:101359. doi: 10.1016/j.smrv.2020.101359. Epub 2020 Jul 10. PMID 32805557
- [Background] Srivanitchapoom P, Pandey S, Hallett M. Restless legs syndrome and pregnancy: a review. Parkinsonism Relat Disord. 2014 Jul;20(7):716-22. doi: 10.1016/j.parkreldis.2014.03.027. Epub 2014 Apr 8. PMID 24768121
- [Background] Silber MH, Buchfuhrer MJ, Earley CJ, Koo BB, Manconi M, Winkelman JW; Scientific and Medical Advisory Board of the Restless Legs Syndrome Foundation. The Management of Restless Legs Syndrome: An Updated Algorithm. Mayo Clin Proc. 2021 Jul;96(7):1921-1937. doi: 10.1016/j.mayocp.2020.12.026. PMID 34218864
- [Background] Sawatari H, Yoshimura C, Amagase H, Takewaka M, Nakashima K, Imaoka C, Obama H, Miyanaga N, Ando SI. Relationship between Restless legs syndrome associated symptoms and presence of depression during pregnancy. Women Health. 2022 Mar;62(3):265-271. doi: 10.1080/03630242.2022.2055698. Epub 2022 Mar 30. PMID 35354362
- [Background] Salehi-Pourmehr H, Atayi M, Mahdavi N, Aletaha R, Kashtkar M, Sharifimoghadam S, Hassanzadeh R, Hajebrahimi S. Is sacral neuromodulation effective and safe in pregnancy? A systematic review. Neurourol Urodyn. 2023 Aug;42(6):1329-1343. doi: 10.1002/nau.25224. Epub 2023 Jun 8. PMID 37288591
- [Background] Roy A, Ojile J, Kram J, Olin J, Rosenberg R, Hudson JD, Bogan RK, Charlesworth JD. Long-term efficacy and safety of tonic motor activation for treatment of medication-refractory restless legs syndrome: A 24-Week Open-Label Extension Study. Sleep. 2023 Oct 11;46(10):zsad188. doi: 10.1093/sleep/zsad188. PMID 37439365
- [Background] Rosen H, Yogev Y. Assessment of uterine contractions in labor and delivery. Am J Obstet Gynecol. 2023 May;228(5S):S1209-S1221. doi: 10.1016/j.ajog.2022.09.003. Epub 2023 Mar 19. PMID 37164494
- [Background] Ozer I, Guzel I, Orhan G, Erkilinc S, Oztekin N, Ak F, Tasci Y. A prospective case control questionnaire study for restless leg syndrome on 600 pregnant women. J Matern Fetal Neonatal Med. 2017 Dec;30(24):2895-2899. doi: 10.3109/14767058.2016.1170801. Epub 2017 Apr 21. PMID 27019150
- [Background] Ramirez JO, Cabrera SA, Hidalgo H, Cabrera SG, Linnebank M, Bassetti CL, Kallweit U. Is preeclampsia associated with restless legs syndrome? Sleep Med. 2013 Sep;14(9):894-6. doi: 10.1016/j.sleep.2013.03.013. Epub 2013 Jul 23. PMID 23891236
- [Background] Liu G, Li L, Zhang J, Xue R, Zhao X, Zhu K, Wang Y, Xiao L, Shangguan J. Restless legs syndrome and pregnancy or delivery complications in China: a representative survey. Sleep Med. 2016 Jan;17:158-62. doi: 10.1016/j.sleep.2015.02.541. Epub 2015 May 4. PMID 26847992
- [Background] Miller MA, Mehta N, Clark-Bilodeau C, Bourjeily G. Sleep Pharmacotherapy for Common Sleep Disorders in Pregnancy and Lactation. Chest. 2020 Jan;157(1):184-197. doi: 10.1016/j.chest.2019.09.026. Epub 2019 Oct 14. PMID 31622589
- [Background] Katsura D, Tsuji S, Hayashi K, Tokoro S, Hoshiyama T, Kita N, Murakami T. Maternal and foetal physiological response of sacral surface electrical stimulation during pregnancy: A preliminary study. Exp Physiol. 2022 May;107(5):508-514. doi: 10.1113/EP090187. Epub 2022 Apr 3. PMID 35293045
- [Background] Jia YJ, Ghi T, Pereira S, Gracia Perez-Bonfils A, Chandraharan E. Pathophysiological interpretation of fetal heart rate tracings in clinical practice. Am J Obstet Gynecol. 2023 Jun;228(6):622-644. doi: 10.1016/j.ajog.2022.05.023. PMID 37270259
- [Background] Jahani Kondori M, Kolla BP, Moore KM, Mansukhani MP. Management of Restless Legs Syndrome in Pregnancy and Lactation. J Prim Care Community Health. 2020 Jan-Dec;11:2150132720905950. doi: 10.1177/2150132720905950. PMID 32054396
- [Background] Harrison EG, Keating JL, Morgan PE. Non-pharmacological interventions for restless legs syndrome: a systematic review of randomised controlled trials. Disabil Rehabil. 2019 Aug;41(17):2006-2014. doi: 10.1080/09638288.2018.1453875. Epub 2018 Mar 21. PMID 29561180
- [Background] Frenken MWE, van der Woude DAA, Dieleman JP, Oei SG, van Laar JOEH. The association between uterine contraction frequency and fetal scalp pH in women with suspicious or pathological fetal heart rate tracings: A retrospective study. Eur J Obstet Gynecol Reprod Biol. 2022 Apr;271:1-6. doi: 10.1016/j.ejogrb.2022.01.023. Epub 2022 Feb 1. PMID 35131629
- [Background] Evans MI, Britt DW, Worth J, Mussalli G, Evans SM, Devoe LD. Uterine contraction frequency in the last hour of labor: how many contractions are too many? J Matern Fetal Neonatal Med. 2022 Dec;35(25):8698-8705. doi: 10.1080/14767058.2021.1998893. Epub 2021 Nov 3. PMID 34732091
- [Background] Charlesworth JD, Adlou B, Singh H, Buchfuhrer MJ. Bilateral high-frequency noninvasive peroneal nerve stimulation evokes tonic leg muscle activation for sleep-compatible reduction of restless legs syndrome symptoms. J Clin Sleep Med. 2023 Jul 1;19(7):1199-1209. doi: 10.5664/jcsm.10536. PMID 36856064
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Buchfuhrer MJ, Baker FC, Singh H, Kolotovska V, Adlou B, Anand H, de Zambotti M, Ismail M, Raghunathan S, Charlesworth JD. Noninvasive neuromodulation reduces symptoms of restless legs syndrome. J Clin Sleep Med. 2021 Aug 1;17(8):1685-1694. doi: 10.5664/jcsm.9404. PMID 33949942
- [Background] Bogan RK, Roy A, Kram J, Ojile J, Rosenberg R, Hudson JD, Scheuller HS, Winkelman JW, Charlesworth JD. Efficacy and safety of tonic motor activation (TOMAC) for medication-refractory restless legs syndrome: a randomized clinical trial. Sleep. 2023 Oct 11;46(10):zsad190. doi: 10.1093/sleep/zsad190. PMID 37458698
- [Background] Arnold JJ, Gawrys BL. Intrapartum Fetal Monitoring. Am Fam Physician. 2020 Aug 1;102(3):158-167. PMID 32735438